CLINICAL TRIAL: NCT00537641
Title: Prevalence and Severity of Nocturnal Oxygenation and Ventilation Failure in Patients With Amyotrophic Lateral Sclerosis Using Noninvasive Ventilation
Brief Title: Efficacy of Noninvasive Ventilation in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAC2000
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: noninvasive ventilation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will test the hypothesis that noninvasive ventilation (NIV) as prescribed in current medical practice for use in amyotrophic Lateral Sclerosis (ALS) patients fails to deliver adequate breathing support over a night of use in the patient's home. ALS patients who come to the ALS Center for their routine 3 month follow up exam and are currently using NIV will be asked to complete questionnaires regarding their quality of sleep, quality of life and general level of function, and to undergo a home sleep study, using a safe, comfortable and reliable breathing monitoring system during a night of sleep. If the questionnaires or the sleep study show failure of the breathing device, the investigators will work with the patient to fix the problem and then offer a second study to make sure that the changes were helpful. The results of this study may help to develop subsequent studies and to improve the guidelines used for care of ALS patients.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS), also known as "Lou Gehrig's Disease", is a fatal disorder that causes breathing failure due to progressive weakness of the muscles of breathing. Breathing assist devices known as noninvasive ventilation (NIV) are offered to ALS patients when their breathing function worsens. These devices deliver breathing assistance via a mask on the nose or nose and mouth, and are thought to be particularly important to be used during sleep, when breathing often becomes more shallow and irregular. However, although these devices have become the standard of therapy in ALS patients once their lung function worsens, it remains unclear how effective these devices actually are when a patient is sleeping, partly because of the practical difficulties in applying the device properly and keeping it applied throughout the sleep period, and partly because they are most commonly prescribed without objective evidence regarding how much breathing support the patient needs as the disease progresses and the breathing muscles weaken further.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of amyotrophic lateral sclerosis (El Escorial criteria)
* age 18 to 18 years old
* using nocturnal noninvasive ventilation to treat respiratory insufficiency at least 4 hours per night, for at least 4 nights per week

Exclusion Criteria:

* inability to safely use NIPPV because of bulbar dysfunction
* indications for tracheostomy assisted ventilation due to inability to clear secretions from the airway
* presence of comorbid conditions with a life expectancy < 6 months
* presence of advanced dementia
* unwillingness to follow up at the Eleanor and Lou Gehrig ALS/MDA Center at Columbia University on a regular basis
* previously diagnosed obstructive sleep apnea
* residence outside the New York metropolitan area.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALS who are using nocturnal noninvasive ventilation to treat respiratory insufficiency will be screened for eligibility as below.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Tolerance of bilevel PAP | Up to 3 months
  The ALS Functional Rating Scale - Revised (ALSFRS-R) will be administered to measure tolerance.
Score on Epworth Sleepiness Scale | Up to 3 months
  Objective evidence of nocturnal sleep-disordered breathing on the bilevel PAP will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Basner, MD, Principal Investigator — Columbia University
Locations (1):
- Eleanor and Lou Gehrig ALS/MDA Center at Columbia University, New York, New York, United States